CLINICAL TRIAL: NCT00527085
Title: A Multicenter, Randomized, Placebo-controlled, Double-blind, 12-month Study to Assess the Effects of an Oral Calcimimetic Agent (AMG 073) on Renal Osteodystrophy in Hemodialysis Patients With Secondary Hyperparathyroidism
Brief Title: 12-month Study of AMG 073 in Renal Osteodystrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20010141
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Renal Osteodystrophy
MeSH Terms: conditions — Chronic Kidney Disease-Mineral and Bone Disorder | interventions — Cinacalcet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- AMG 073 (Experimental)
  Interventions: Drug: AMG 073
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMG 073 — 30 mg QD orally 50 mg QD orally 70 mg QD orally 90 mg QD orally 120 mg QD orally 180 mg QD orally
  Arms: AMG 073
Drug: Placebo — 30 mg QD orally 50 mg QD orally 70 mg QD orally 90 mg QD orally 120 mg QD orally 180 mg QD orally
  Arms: Placebo

SUMMARY:
4 doses of AMG 073 or placebo over 52 weeks after a 30-day screening period. Throughout the study, labs will be drawn to measure analytes such as iPTH and corrected calcium. In addition, a bone biopsy will be performed at screening and at the end of study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age of greater
* Using effective contraceptive measures
* iPTH greater than or equal to 300 pg/mL
* Serum Calcium greater than or equal to 8.4 mg/dL; Hemoglobin greater than 9
* Stable hemodialysis for 1 month prior to day 1

Exclusion Criteria:

* Any unstable medical condition
* Pregnant or nursing women Recent parathyroidectomy
* Change in Vitamin D therapy
* Recent MI, Seizure, Malignancy, GI Disorder
* Inability to swallow tablets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2001-10; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of AMG 073 compared with placebo on renal osteodystrophy as assessed by bone histomorphometry | entire study

SECONDARY OUTCOMES:
To evaluate the effects of AMG 073 compared with placebo on intact parathyroid hormone (iPTH), bone-specific alkaline phosphatase (BALP), serum N-Telopeptide (N-Tx), and calcium x phosphorus product concentrations | entire study
To evaluate the feasibility of measuring physical activity with accelerometry | entire study
To evaluate the safety and tolerability of AMG 073 compared with placebo | entire study

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Malluche HH, Monier-Faugere MC, Wang G, Fraza O JM, Charytan C, Coburn JW, Coyne DW, Kaplan MR, Baker N, McCary LC, Turner SA, Goodman WG. An assessment of cinacalcet HCl effects on bone histology in dialysis patients with secondary hyperparathyroidism. Clin Nephrol. 2008 Apr;69(4):269-78. doi: 10.5414/cnp69269. PMID 18397701
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_38_AMG_073_20010141.pdf
- See also: FDA-approved Drug Labeling — http://www.sensipar.com/
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com